CLINICAL TRIAL: NCT03372213
Title: Dietary Quality by At-home and Away-from-home Food Sources in the Supplemental Nutrition Assistance Program (SNAP)
Brief Title: Healthfulness of Food From Grocery Stores Versus Eating Out Among People Receiving Food Benefits (SNAP)
Acronym: SNAP
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 12-2163; R01DK098072 (NIH); P2CHD050924 (NIH)
Record Dates: First submitted 2017-12-01; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 2003-2004: Adults 20-64 at or below 130% of the federal poverty level who completed one 24-hour dietary recall
- 2005-2006: Adults 20-64 at or below 130% of the federal poverty level who completed one 24-hour dietary recall
- 2011-2012: Adults 20-64 at or below 130% of the federal poverty level who completed one 24-hour dietary recall
- 2013-2014: Adults 20-64 at or below 130% of the federal poverty level who completed one 24-hour dietary recall

SUMMARY:
The objective of this cross-sectional study was to characterize the dietary intake of SNAP participants and nonparticipants by food source, including grocery stores, sit-down restaurants, and fast food.

DETAILED DESCRIPTION:
The study used 4,237 low-income adults from the National Health and Nutrition Examination Survey (NHANES) (2003-2006 and 2011-2014). De-identified data was collected from demographic questionnaires and 24 hour dietary recalls. We assessed intake of calories, solid fats, added sugars, and servings of non-starchy vegetables, whole fruits, and whole grains, by food source in SNAP participants and income-eligible nonparticipants. Associations between SNAP participation and dietary intake were analyzed using multivariate linear regression controlling for relevant sociodemographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 20 - 64
* At or below 200% of the federal poverty level
* Completed at least one 24-hour dietary recall

Exclusion Criteria:

* Younger than 20 years old or 65 years and older
* Income above 200% the federal poverty level
* No participation in dietary recall

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 4,237 low-income adults in the National Health and Nutrition Examination Survey (NHANES) (2003-2006 and 2011-2014)
Sampling Method: Probability Sample
Enrollment: 4237 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Caloric intake | 2003-2014
  Number of calories consumed by SNAP participants compared to nonparticipants in 2003-2006 and 2011-2014 by source of food (including grocery stores, fast food restaurants, sit-down restaurants and other sources). SNAP participants will be compared to income-eligible nonparticipants at income levels up to 200% of the federal poverty level.
Solid fat | 2003-2014
  Number of grams of solid fat and percent of intake from solid fat consumed by SNAP participants compared to nonparticipants in 2003-2006 and 2011-2014 by source of food (including grocery stores, fast food restaurants, sit-down restaurants and other sources). SNAP participants will be compared to income-eligible nonparticipants at income levels up to 200% of the federal poverty level.
Added sugar | 2003-2014
  Number of grams of added sugar and percent of intake from added sugar consumed by SNAP participants compared to nonparticipants in 2003-2006 and 2011-2014 by source of food (including grocery stores, fast food restaurants, sit-down restaurants and other sources). SNAP participants will be compared to income-eligible nonparticipants at income levels up to 200% of the federal poverty level.
Non-starchy vegetables | 2003-2014
  Cup-equivalent servings of non-starchy vegetables consumed by SNAP participants compared to nonparticipants in 2003-2006 and 2011-2014 by source of food (including grocery stores, fast food restaurants, sit-down restaurants and other sources). SNAP participants will be compared to income-eligible nonparticipants at income levels up to 200% of the federal poverty level.
Whole fruit | 2003-2014
  Cup-equivalent servings of whole fruits consumed by SNAP participants compared to nonparticipants in 2003-2006 and 2011-2014 by source of food (including grocery stores, fast food restaurants, sit-down restaurants and other sources). SNAP participants will be compared to income-eligible nonparticipants at income levels up to 200% of the federal poverty level.
Whole grains | 2003-2014
  Ounce-equivalents of whole grains consumed by SNAP participants compared to nonparticipants in 2003-2006 and 2011-2014 by source of food (including grocery stores, fast food restaurants, sit-down restaurants and other sources). SNAP participants will be compared to income-eligible nonparticipants at income levels up to 200% of the federal poverty level.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Popkin, PhD, Principal Investigator — University of North Carolina, Chapel Hill